CLINICAL TRIAL: NCT03569111
Title: Clinical Description of a Bronchoscopic Approach to Ablate Lung Nodules Using the Emprint™ Ablation Catheter Kit With Thermosphere™ Technology
Brief Title: Clinical Description of a Bronchoscopic Approach to Ablate Lung Nodules Using the Emprint™ Ablation Catheter
Acronym: NAVABLATE
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT18010ILSBA
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-04

CONDITIONS: Cancer, Lung; Cancer, Metastatic to Lung
Keywords: Lung Nodule; Bronchoscopy; Ablation, Microwave
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bronchoscopic ablation catheter — The Emprint™ Ablation Catheter Kit with Thermosphere™ Technology is deployed endoscopically and will be used to conduct bronchoscopic ablations in the lung using the superDimension™ navigation system.

SUMMARY:
The purpose of this investigation is to characterize the safety and performance of the Emprint™ Ablation Catheter Kit with Thermosphere™ Technology in clinical use.

This is a prospective, single-arm, multicenter, non-randomized study. Up to 3 sites in up to 3 countries will enroll up to 30 subjects in total. The study is designed to characterize the safety and performance of the bronchoscopic ablation procedure using the Emprint™ Ablation Catheter Kit with Thermosphere™ Technology.

DETAILED DESCRIPTION:
The primary objective of this prospective, single-arm, multicenter, non-randomized study is to characterize the safety of the Emprint™ Ablation Catheter Kit with Thermosphere™ Technology device in subjects undergoing lung ablation procedures.

The primary endpoint is the composite rate of adverse events related to the Emprint™ Ablation Catheter Kit with Thermosphere™ Technology through 1-month follow-up.

The following secondary endpoints will be evaluated:

* Composite rate of serious adverse events related to the Emprint™ Ablation Catheter Kit with Thermosphere™ Technology through 1-month follow-up.
* Composite rate of all adverse events related to the procedure or study devices through 1-month follow-up.
* Composite rate of all serious adverse events related to the procedure or study devices through 1-month follow-up.
* Patient satisfaction and pain (Bronchoscopic Ablation Patient Pain and Satisfaction Survey)
* Quality of life (EQ-5D Scale)
* Technical success
* Technique efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject has provided informed consent
3. Subject is able and willing to comply with the study follow-up schedule
4. Subject has a definitive diagnosis of cancer in the lung
5. Target nodule is ≤ 30mm in maximum diameter
6. There is ≥ 5mm of nodule-free lung parenchyma between target nodule and pleura or fissure
7. Subject is a candidate for an elective electromagnetic navigation bronchoscopy (ENB) procedure
8. Subject is a candidate for an elective lung ablation procedure according to standard of care and product Instructions for Use
9. Subject is not a candidate for lung surgery or refuses lung surgery
10. Subject is not a candidate for stereotactic body radiation therapy (SBRT) or refuses SBRT

Exclusion Criteria:

1. Target nodule is abutting main stem bronchus, main pulmonary vasculature, esophagus and/or trachea
2. Patients currently diagnosed with Global Initiative for Chronic Obstructive Lung Disease (GOLD) Stage IV emphysema
3. Female subjects who are pregnant or nursing as determined by standard site practices
4. Subject has participated in an investigational drug or device research study within 30 days of enrollment that would interfere with this study
5. The investigator determines that participation in the study may jeopardize the safety or welfare of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included must have a cancerous lung nodule, and will be candidates for an elective ENB and lung ablation procedure. Subjects themselves will need to provide written consent and agree to attend study visits and complete questionnaires. Up to 30 subjects will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lau, MA DPhil FRCS(CTh), Principal Investigator — St Bartholomew's Hosptial
Locations (2):
- Prince of Wales Hospital, Hong Kong, Hong Kong
- St. Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NAVABLATE (Single-arm Study): Observational NAVABLATE arm (single-arm, no comparator)
Period: Overall Study
Arm/Group | NAVABLATE (Single-arm Study)
Started | 30
Procedure | 30
1-Month | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 30 subjects were enrolled. The bronchoscopic ablation procedure was performed on 1 lesion for each subject.
Units Other Than Participants: Lesions
Groups:
- NAVABLATE (Single-arm Study): Observational NAVABLATE arm (single-arm study, no comparator)
Arm/Group | NAVABLATE (Single-arm Study)
Number analyzed (Participants) | 30
Number analyzed (Lesions) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 14
  United Kingdom | 16
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 10
Tobacco use (current or former) [Count of Participants; unit: Participants] | 20
Prior lung procedures performed [Count of Participants; unit: Participants] — Subjects could have more than one prior lung procedure performed.
  Participants
    Lung surgery | 11
    Radiotherapy | 1
    Non-surgical biopsy procedure | 19
No prior lung procedure performed [Count of Participants; unit: Participants] | 7
Eligibility for Lung surgery or SBRT [Count of Participants; unit: Participants]
  Not a candidate for lung surgery or Stereotactic body radiation therapy (SBRT) | 14
  Declined both lung surgery and SBRT | 10
  Not a candidate for lung surgery and declined SBRT | 5
  Not a candidate for SBRT and declined lung surgery | 1
State of cancer diagnosis [Count of Participants; unit: Participants]
  Primary Lung Cancer | 20
  Oligometastatic | 10
Nodule size (mm) [Mean (Standard Deviation); unit: millimeters] — Nodule size from pre-procedure CT scan
  millimeters | 13.7 (5.3)
Lobe zone of nodule [Count of Units; unit: Lesions]
  Peripheral third of lung | 19
  Middle third of lung | 11
  Proximal third of lung | 0
Lobe location [Count of Participants; unit: Participants]
  Right Upper Lobe | 10
  Right Middle Lobe | 2
  Right Lower Lobe | 8
  Left Upper Lobe | 6
  Left Lower Lobe | 4
Bronchus sign present [Count of Participants; unit: Participants] — Bronchus sign present based on pre-procedure CT scan
  Participants | 14
Lesion morphology [Count of Units; unit: Lesions]
  Suzuki class 1 or 2 (Pure Ground Glass Opacity [GGO] or Mostly GGO) | 3
  Suzuki class 3 or 4 (Halo or Mixed) | 5
  Suzuki class 5 or 6 (Solid Pattern with GGO or Solid) | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With AEs Related to the Emprint™ Ablation Catheter Kit With Thermosphere™ Technology
Description: The primary endpoint is the rate of adverse events (AEs) related to the Emprint™ Ablation Catheter Kit with Thermosphere™ Technology through 1-month follow-up.
Time Frame: During procedure through 1-month follow-up (an average of 20-40 days post-procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | NAVABLATE (Single-Arm Study)
Number analyzed (Participants) | 30
Participants | 1

2. Secondary Outcome: Number of Participants With SAEs Related to the Emprint™ Ablation Catheter Kit With Thermosphere™ Technology
Description: Rate of serious AEs (SAEs) related to the Emprint™ Ablation Catheter Kit with Thermosphere™ Technology through 1-month follow-up.
Time Frame: During procedure through 1-month follow-up (an average of 20-40 days post-procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | NAVABLATE (Single-arm Study)
Number analyzed (Participants) | 30
Participants | 0

3. Secondary Outcome: Number of Participants With AEs Related to Study Procedure or Study Devices
Description: Rate of all AEs related to the procedure or study devices through 1-month follow-up.
  Rate of all AEs related to the procedure or study devices through 1-month follow-up was also measured based on Common Terminology Criteria for Adverse Events (CTCAE) classification. CTCAE grading is evaluated on a scale from 1-5 (1 - mild; intervention not indicated; 5 - most severe; death related to AE). Subjects could have more than one AE with different CTCAE Grades.
Time Frame: During procedure through 1-month follow-up (an average of 20-40 days post-procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | NAVABLATE (Single-arm Study)
Number analyzed (Participants) | 30
Participants
  Composite rate of all AEs related to the procedure or study devices | 21
  CTCAE Grade 1 | 15
  CTCAE Grade 2 | 11
  CTCAE Grade 3 | 4
  CTCAE Grade 4 | 0
  CTCAE Grade 5 | 0

4. Secondary Outcome: Number of Participants With SAEs Related to the Study Procedure or Study Devices
Description: Rate of all SAEs related to the procedure or study devices through 1-month follow-up.
Time Frame: During procedure through 1-month follow-up (an average of 20-40 days post-procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | NAVABLATE (Single-arm Study)
Number analyzed (Participants) | 30
Participants | 4

5. Secondary Outcome: Score of Patient Satisfaction, Pain, and Breathlessness
Description: Patient satisfaction, pain, and breathlessness (Bronchoscopic Ablation Patient Pain and Satisfaction Survey)
  At the 1-month visit, subjects assessed their pain/discomfort and breathlessness based on how they recall feeling at 3 different timepoints. The timepoints were immediately, one week, and one month after the bronchoscopic ablation procedure. Pain or discomfort were evaluated on a scale from 0-10 (10 - severe/interferes with basic needs). Breathlessness was evaluated on a scale from 1-5 (5 - too breathless to leave the house, or breathless when undressing).
  Subjects also evaluated their willingness to have the procedure performed again on a scale from 1-5 (5 - extremely likely), how likely they would recommend the procedure to family and friends on a scale from 1-5 (5 - extremely likely), and how satisfied they were with the procedure on a scale from 1-5 (5 - extremely satisfied).
Time Frame: Immediately following the procedure, 1 week post-procedure, 1-month post-procedure; all were collected at the 1-month follow-up visit (20-40 days post-procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAVABLATE (Single-arm Study)
Number analyzed (Participants) | 30
score on a scale
  Pain/discomfort immediately after procedure | 1.5 (2.2)
  Pain/discomfort one week after procedure | 1.4 (1.8)
  Pain/discomfort one month after procedure | 0.5 (1.1)
  Breathlessness immediately after procedure | 1.8 (1.0)
  Breathlessness one week after procedure | 1.6 (1.0)
  Breathlessness one month after procedure | 1.5 (0.9)
  Willingness to have the procedure performed again | 4.8 (0.8)
  Likelihood to recommend the procedure to family and friends | 4.9 (0.4)
  Satisfaction with procedure at 1-month | 4.8 (0.4)

6. Secondary Outcome: Score of Current Health State From Quality of Life Survey
Description: Quality of life evaluation based on EuroQol [EQ-5D-3L] survey. The questions from the survey surround current health status. The subjects assessed their current health state on a scale of 0-100 (100 being the best health state imaginable).
Time Frame: Baseline and 1-month
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAVABLATE (Single-arm Study)
Number analyzed (Participants) | 30
score on a scale
  Baseline | 74.6 (12.8)
  1-month | 77.4 (14.2)

7. Secondary Outcome: Number of Lung Nodules Evaluated as Being Treated According to the Study Protocol
Description: Technical success: An evaluation of whether the lung nodule was treated according to the study protocol as determined at the immediate post-procedural timepoint. This is in contrast to procedures in which the protocol could not be executed completely, either for technical reasons or for reasons related to comorbid disease.
Time Frame: Immediately post-procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Units; unit: lesions ablated
Units Other Than Participants: lesions ablated
Arm/Group | NAVABLATE (Single-arm Study)
Number analyzed (Participants) | 30
Number analyzed (lesions ablated) | 30
lesions ablated | 30

8. Secondary Outcome: Number of Lung Nodules Evaluated as Being Effectively Ablated
Description: Technique efficacy: An evaluation of whether the lung nodule was effectively ablated. Evaluates whether complete ablation of the nodule was achieved as evidenced by CT imaging follow-up 1-month post-procedure (including a window of 20-40 days post-procedure).
Time Frame: 1-month follow-up (an average of 20-40 days post-procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Units; unit: lesions ablated
Units Other Than Participants: lesions ablated
Arm/Group | NAVABLATE (Single-arm Study)
Number analyzed (Participants) | 30
Number analyzed (lesions ablated) | 30
lesions ablated | 30

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the point of enrollment (when the Emprint catheter was inserted into the compatible extended working channel) up to 1-month post-procedure.
Description: Adverse event definitions were based on ISO 14155:2011. All AEs related to the Emprint™ Ablation Catheter Kit with Thermosphere™ Technology, accessory devices, or study procedures were required to be reported.
Arm/Group | NAVABLATE (Single-arm Study)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVABLATE (Single-arm Study) (N=30)
Administration site infection (Infections and infestations) | 1 (1)
Post ablation syndrome (Injury, poisoning and procedural complications) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVABLATE (Single-arm Study) (N=30)
Bradycardia (Cardiac disorders) | 1 (1)
Chest discomfort (General disorders) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Post ablation syndrome (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 13 (15)
Unwanted awareness during anaesthesia (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator shall not publish the Study results until after Sponsor's multi-site publication and final study results are complete or until the elapse of twelve (12) months from the close of the Study at all Study sites, whichever occurs first; unless approved by Sponsor.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03569111/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03569111/SAP_001.pdf